CLINICAL TRIAL: NCT03799146
Title: A Randomized Controlled Trial to Identify the Effect and the Working Mechanisms of MyPlan 2.0, a Self-regulation-based e- and mHealth Intervention Targeting Physical Activity and Sedentary Behaviour, in Older Adults
Brief Title: Identifying the Effect and Working Mechanisms of MyPlan 2.0 in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MyPlan2.0_older_adults_50
Record Dates: First submitted 2019-01-07; First posted 2019-01-10 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Overweight
Keywords: physical activity; sedentary behaviour; eHealth; mHealth; self-regulation; behaviour change techniques
MeSH Terms: conditions — Overweight; Motor Activity; Self-Control | interventions — Waiting Lists

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with two groups: intervention group and waiting-list control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants will receive the e- and mHealth intervention 'MyPlan 2.0'.
  Interventions: Behavioral: MyPlan 2.0
- Waiting List control group (Experimental): Participants will not receive the e- and mHealth intervention 'MyPlan 2.0', but will be given access to the intervention after all testing phases.
  Interventions: Other: Waiting List

INTERVENTIONS:
Behavioral: MyPlan 2.0 — MyPlan 2.0 consists of five sessions. During these five sessions the following behaviour change techniques are used to motivate users to be more physically active or to sit less: exploring risk perceptions and perceived benefits, exploring social support, providing feedback, action planning, coping planning and monitoring.
  Arms: Intervention group
Other: Waiting List — Waiting List control group
  Arms: Waiting List control group

SUMMARY:
The aim of this study is to investigate whether and how 'MyPlan 2.0' helps older adults to be more physically active or less sedentary. Two groups will be created, an intervention group and a waiting-list control group.

DETAILED DESCRIPTION:
The aim of this study is to investigate whether and how 'MyPlan 2.0' helps older adults to be more physically active or less sedentary. Two groups will be created, an intervention group and a waiting-list control group. Both groups will be tested during three testing waves: pretest, posttest and follow-up test. Only the intervention group will be given acces to 'MyPlan 2.0'.

'MyPlan 2.0' consists of a website and mobile application targeting physical activity and sedentary behaviour. The intervention has a duration of five weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have access to internet
* Being computer literate

Exclusion Criteria:

* non Dutch speaking

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Change in objective total, light and moderate-to-vigorous physical activity (PA) | Pretest, posttest (6 weeks) and follow-up (6 months)
  Change in amount of total, light and moderate-to-vigorous physical activity, measured via accelerometers
Change in objective sedentary behaviour | Pretest, posttest (6 weeks) and follow-up (6 months)
  Change in amount of total sitting time, measured via accelerometers
Change in self-reported total, moderate and moderate-to-vigorous physical activity (PA) as well as total work-related, transport-related, household-related and leisure time PA. | Pretest, posttest (6 weeks) and follow-up (6 months)
  Change in amount of total, light and moderate-to-vigorous PA well as total work-related, transport-related, household-related and leisure time PA will be measured via the International Physical Activity Questionnaire (IPAQ). The IPAQ measures physical activity in four domains: work, transport, household and leisure time. Higher scores indicate higher levels of physical activity. For each scale the minimum value is 0. We will use the method described by Dubuy et al. (2013) to truncate the data.
Change in self-reported sedentary behaviour | Pretest, posttest (6 weeks) and follow-up (6 months)
  Change in amount of total sitting time, measured via the LASA sedentary behaviour self-report questionnaire. The total score is calculated by summing all 10 items.The minimum value is 0 and the maximum value is 24 hours. However, data will be truncated at 16 hours.

SECONDARY OUTCOMES:
Change in self-efficacy | Pretest, after week 1, after week 2, after week 3, after week 4, posttest (6 weeks), and follow-up (6 months)
  Change in amount of self-efficacy to change behaviour, measured via 5 validated items (questionnaire). These items were created by the involved research groups. For each item, the scale ranges from 1 to 10. The average score on the five items will be considered the final score.
Change in outcome expectancies | Pretest, after week 1, after week 2, after week 3, after week 4, posttest (6 weeks), and follow-up (6 months
  Outcome expectancies regarding the behaviour change, measured via 5 validated items (questionnaire). These items were created by the involved research groups. For each item, the scale ranges from 1 to 10. The average score on the five items will be considered the final score.
Change in risk perception | Pretest, after week 1, after week 2, after week 3, after week 4, posttest (6 weeks), and follow-up (6 months
  Risk perception about the behaviour, measured via 4 validated items (questionnaire). These items were created by the involved research groups. For each item, the scale ranges from 1 to 10. The average score on the four items will be considered the final score
Change in intention | Pretest, after week 1, after week 2, after week 3, after week 4, posttest (6 weeks), and follow-up (6 months
  Amount of intention to change the behaviour, measured via 3 validated items (questionnaire). These items were created by the involved research groups. For each item, the scale ranges from 1 to 10. The average score on the three items will be considered the final score.
Change in action planning | Pretest, after week 1, after week 2, after week 3, after week 4, posttest (6 weeks), and follow-up (6 months
  Amount of action planning for behaviour change, measured via 3 validated items (questionnaire). These items were created by the involved research groups. For each item, the scale ranges from 1 to 10. The average score on the three items will be considered the final score.
Change in coping planning | Pretest, after week 1, after week 2, after week 3, after week 4, posttest (6 weeks), and follow-up (6 months
  Amount of coping planning for behaviour change, measured via 3 validated items (questionnaire). These items were created by the involved research groups. For each item, the scale ranges from 1 to 10. The average score on the three items will be considered the final score.

CONTACTS AND LOCATIONS:
Overall Officials: Ilse De Bourdeaudhuij, Principal Investigator — University Ghent; Geert Crombez, Principal Investigator — University Ghent
Locations (1):
- Department of Movement and Sports Sciences, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Poppe L, De Bourdeaudhuij I, Verloigne M, Shadid S, Van Cauwenberg J, Compernolle S, Crombez G. Efficacy of a Self-Regulation-Based Electronic and Mobile Health Intervention Targeting an Active Lifestyle in Adults Having Type 2 Diabetes and in Adults Aged 50 Years or Older: Two Randomized Controlled Trials. J Med Internet Res. 2019 Aug 2;21(8):e13363. doi: 10.2196/13363. PMID 31376274